CLINICAL TRIAL: NCT01749384
Title: Phase I Study of Tivantinib Plus Bevacizumab
Brief Title: Tivantinib and Bevacizumab in Treating Patients With Solid Tumors That Are Metastatic or Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02765; NCI-2012-02765 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UPCI 12-085; UPCI# 12-085; 9153 (Other: University of Pittsburgh Cancer Institute (UPCI)); 9153 (Other: CTEP); P30CA047904 (NIH); U01CA099168 (NIH); UM1CA186690 (NIH)
Record Dates: First submitted 2012-12-11; First posted 2012-12-13 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Solid Neoplasm
MeSH Terms: interventions — Bevacizumab; Immunoglobulin G; Disulfides; ARQ 197

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (bevacizumab, tivantinib) (Experimental): Patients receive bevacizumab IV over 30-90 minutes on days -15, 1, and 15 (day -15 of course 1 only) and tivantinib PO BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Tivantinib

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar FKB238; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Tivantinib — Given PO
  Other Names: ARQ 197; ARQ-197; c-Met Inhibitor ARQ 197

SUMMARY:
This phase I trial studies the side effects of and best dose of tivantinib when given together with bevacizumab in treating patients with solid tumors that have spread to other areas of the body or cannot be removed by surgery. Tivantinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as bevacizumab, may block tumor growth in different ways by targeting certain cells. Bevacizumab may also stop the growth of cancer by blocking blood flow to the tumor. Giving tivantinib together with bevacizumab may work better in treating tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the recommended phase II dose (RP2D) of the vascular endothelial growth factor (VEGF) monoclonal antibody, bevacizumab in combination with the allosteric met proto-oncogene (MET) inhibitor, tivantinib, in patients with advanced solid tumors.

SECONDARY OBJECTIVES:

I. Describe the dose-limiting toxicity (DLT) and other toxicities associated with bevacizumab in combination with tivantinib as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version (v) 4.0.

II. Document anti-tumor activity of bevacizumab in combination with tivantinib in patients with advanced solid tumors.

III. Determine the pharmacokinetics of tivantinib when administered in combination with bevacizumab in patients with advanced solid tumors.

IV. Perform cytochrome P450 family 2, subfamily C, polypeptide 19 (CYP2C19) genotyping on all subjects and correlate with pharmacokinetics and toxicity.

V. Assess the effect of bevacizumab plus tivantinib on plasma components of the hepatocellular growth factor (HGF)-MET signaling pathway (HGF, HGF activator [HGFA]) and VEGF signaling pathway (VEGF A, B, C, D and placental growth factor [PIGF]).

VI. Assess tissue (tumor and skin) protein biomarkers before and after study treatment including MET, phospho-MET^tyrosine (Tyr)1349 and phosphor-focal adhesion kinase (FAK)^Tyr861.

VII. Assess early therapy response by quantitative biomarker imaging fludeoxyglucose F 18 (F-18 FDG) positron emission tomography (PET) and magnetic imaging resonance (MRI) on a smaller sample (n up to 15) of subjects willing to participate in the imaging assessment through UPCI 12-096.

OUTLINE: This is a dose-escalation study of tivantinib.

Patients receive bevacizumab intravenously (IV) over 30-90 minutes on days -15, 1, and 15 (day -15 of course 1 only) and tivantinib orally (PO) twice daily (BID) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed solid tumor malignancy (excluding squamous cell carcinoma of lung) that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
* Patients must have measurable or evaluable disease by Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.1)
* Current diagnosis of type II diabetes mellitus is eligible as long as patient glucose levels are well-controlled (fasting =< 150 mg/dL) with anti-diabetic medication
* Patients must be able to swallow pills and no significant impairment in gastrointestinal absorption
* There are no restrictions on prior therapy:

  * Prior bevacizumab is allowed
  * Prior therapy with inhibitors of MET or HGF is allowed
* Eastern Cooperative Oncology Group (ECOG) performance status must be =< 2 (Karnofsky >= 60%)
* Life expectancy must be greater than 3 months
* Hemoglobin >= 9.0 g/dL
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 X institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional ULN
* Serum or plasma creatinine =< 1.5 X institutional ULN OR creatinine clearance >= 60 mL/min for patients with creatinine levels > 1.5 X institutional ULN
* Urine protein =< +1 on spot urinalysis/urine dipstick; if urine dipstick > +1, a 24-hour urine for protein must be =< 1 G/24 hour (hr)
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of tivantinib administration
* Negative urine or serum pregnancy test within 7 days of start of protocol therapy (for female patients who have not undergone bilateral oophorectomy or hysterectomy)
* Patients must have the ability to understand and the willingness to sign a written informed consent document
* Patients must have available archival tumor tissue (formalin-fixed, paraffin-embedded) for submission of blocks or unstained slides

Exclusion Criteria:

* Patients who have had chemotherapy, monoclonal antibody therapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to start of study drugs or those who have adverse events not resolved to a grade 1 or neuropathy not resolved to =< grade 2 due to agents administered more than 4 weeks earlier
* Major hemorrhagic or thrombotic event within 3 months of start of protocol therapy
* Major surgery within 6 weeks or non-healing wounds
* Patients who have received kinase inhibitor therapy within 2 weeks of start of protocol therapy
* Patients who are receiving any other investigational agents
* Known central nervous system (CNS) disease except for treated brain metastasis; treated brain metastases are defined as having no ongoing requirement for steroids and no evidence of progression or hemorrhage after treatment for at least 3 months, as ascertained by clinical examination and brain imaging (magnetic resonance imaging [MRI] or computed tomography [CT]); (stable dose of non-enzyme-inducing anticonvulsants are allowed); treatment for brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (RS; Gamma Knife, linear accelerator [LINAC], or equivalent) or a combination as deemed appropriate by the treating physician; patients with CNS metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to day 1 will be excluded
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to tivantinib or bevacizumab, or to Chinese hamster ovary cells
* Tivantinib is metabolized by CYP2C19, and to a lesser extent cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4); the metabolism and consequently overall pharmacokinetics of tivantinib could be altered by inhibitors and/or inducers or other substrates of CYP2C19 and CYP3A4; while inhibitors/inducers of these cytochrome P450 isoenzymes are not specifically excluded, investigators should be aware that tivantinib exposure may be altered by the concomitant administration of these drugs; as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, psychiatric illness/social situations that would limit compliance with study requirements
* Patients with clinically significant cardiovascular disease, including any of the following, are excluded:

  * Inadequately controlled hypertension (HTN) (systolic blood pressure [SBP] > 160 mmHg and/or diastolic blood pressure [DBP] > 90 mmHg despite antihypertensive medication)
  * History of cerebrovascular accident (CVA) within 6 months of start of protocol therapy
  * Myocardial infarction or unstable angina within 6 months of start of protocol therapy
  * New York Heart Association grade II or greater congestive heart failure
  * Serious and inadequately controlled cardiac arrhythmia
  * Significant vascular disease (e.g. significant aortic aneurysm, history of aortic dissection)
  * Clinically significant peripheral vascular disease
  * Untreated deep venous thrombosis (DVT) or pulmonary embolism (PE) or DVT/PE which has been treated with therapeutic anticoagulation for less than 6 weeks
* History of hemoptysis in excess of 2.5 mL (1/2 teaspoon ) within 8 weeks prior to first dose of study drug
* Pregnant women are excluded from this study, and breastfeeding should be discontinued if the mother is treated with tivantinib; these potential risks may also apply to bevacizumab
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-12-06 (Actual); Primary Completion 2016-05-24 (Actual); Study Completion 2016-05-24 (Actual)

PRIMARY OUTCOMES:
RP2D of the combination of tivantinib and bevacizumab, defined as the dose level at which the dose-limiting toxicity (DLT) rate is closest to 1/6 graded according to the National Cancer Institute (NCI) CTCAE v4.0 | Up to 28 days

SECONDARY OUTCOMES:
Change in HGF, HGFA, VEGF, and PIGF in plasma by enzyme-linked immunosorbent assay | Baseline to up to day 15 of course 1
  Plasma before and after the treatment will be measured and compared by Wilcoxon signed rank test.
Change in MET, FAK, AKT, STAT3 in skin tissue by immunohistochemistry | Baseline to up to day 15 of course 1
  Skin biomarkers before and after the treatment will be measured and compared by Wilcoxon signed rank test.
Clinical response rate as evaluated by RECIST | Up to 4 weeks after completion of study treatment
  The clinical response rate will be calculated and corresponding 95% exact confidence interval will be provided. The percent changes in tumor sized from the baseline will be presented by the waterfall plot.
Incidence of adverse events graded according to NCI CTCAE v4.0 that are possibly, probably, or definitely related to treatment | Up to 4 weeks after completion of study treatment
  The maximum grade of toxicity for each category of interest will be recorded for each patient and the summary results will be tabulated by category and grade. All DLTs and other serious (grade 3 or greater) toxicity events on a patient-by-patient basis will be described; descriptions will include dose level and any relevant baseline data. Statistics on the number of cycles received by patients and any dose reductions will be tabulated. Toxicity profile for CYP2C19 mutant carriers will be summarized and compared to non-carriers by exact tests when sample size permits.
Pharmacokinetics (PK) of tivantinib when administered in combination with bevacizumab | At days 1, 2, and 15 of course 1
  PK outcomes for CYP2C19 mutant carriers will be summarized and compared to non-carriers by exact tests when sample size permits.

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Appleman, Principal Investigator — University of Pittsburgh Cancer Institute (UPCI)
Locations (2):
- United States (2):
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Maguire WF, Schmitz JC, Scemama J, Czambel K, Lin Y, Green AG, Wu S, Lin H, Puhalla S, Rhee J, Stoller R, Tawbi H, Lee JJ, Wright JJ, Beumer JH, Chu E, Appleman LJ; ETCTN-9153 Study Team. Phase 1 study of safety, pharmacokinetics, and pharmacodynamics of tivantinib in combination with bevacizumab in adult patients with advanced solid tumors. Cancer Chemother Pharmacol. 2021 Oct;88(4):643-654. doi: 10.1007/s00280-021-04317-y. Epub 2021 Jun 23. PMID 34164713